CLINICAL TRIAL: NCT05438147
Title: A Randomized Exploratory Basket Study to Evaluate the Effects of a CT-100 DiNaMo Component on Cognitive Functioning and Mood Symptoms in Adult Participants With a Primary Non-DSM-5 Diagnosis
Brief Title: Effects of a CT-100 DiNaMo Component on Cognitive Functioning and Mood Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Click Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CT-100-D-001
Record Dates: First submitted 2022-06-06; First posted 2022-06-29 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis; Mild Cognitive Impairment; Cancer
Keywords: Digital therapeutics; Phone app; Virtual study
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction; Neoplasms

STUDY DESIGN:
Intervention Model Description: Active Intervention Device vs. Care-as-Usual Control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- CT-100 DiNaMo (Study App) in Patients with Multiple Sclerosis (Active Comparator): Randomized Controlled Study to Evaluate CT-100 DiNaMo (Study App) in Patients with Multiple Sclerosis
  Interventions: Other: CT-100 DiNaMo
- Care-as-Usual control in Patients with Multiple Sclerosis (Sham Comparator): Randomized controlled Study to Evaluate Care-as-Usual control in Patients with Multiple Sclerosis
  Interventions: Other: Care-as-Usual
- CT-100 DiNaMo (Study App) in Patients with Breast or Lung Cancer (Active Comparator): Randomized Controlled Study to Evaluate CT-100 DiNaMo (Study App) in Patients with with Breast or Lung Cancer
  Interventions: Other: CT-100 DiNaMo
- Care-as-Usual control in Patients with Breast or Lung Cancer (Sham Comparator): Randomized Controlled Study to Evaluate Care-as-Usual control in Patients with with Breast or Lung Cancer
  Interventions: Other: Care-as-Usual
- CT-100 DiNaMo (Study App) in Patients with Mild Cognitive Impairment (Active Comparator): Randomized Controlled Study to Evaluate CT-100 DiNaMo (Study App) in Patients with Mild Cognitive Impairment
  Interventions: Other: CT-100 DiNaMo
- Care-as-Usual in Patients with Mild Cognitive Impairment (Sham Comparator): Randomized Controlled Study to Evaluate Care-as-Usual in Patients with Mild Cognitive Impairment
  Interventions: Other: Care-as-Usual

INTERVENTIONS:
Other: CT-100 DiNaMo — Active Treatment (Study App)
  Arms: CT-100 DiNaMo (Study App) in Patients with Breast or Lung Cancer; CT-100 DiNaMo (Study App) in Patients with Mild Cognitive Impairment; CT-100 DiNaMo (Study App) in Patients with Multiple Sclerosis
Other: Care-as-Usual — Care-As-Usual control
  Arms: Care-as-Usual control in Patients with Breast or Lung Cancer; Care-as-Usual control in Patients with Multiple Sclerosis; Care-as-Usual in Patients with Mild Cognitive Impairment

SUMMARY:
CT-100 is a platform that provides an interactive, software based therapeutic component that may be used as part of a multimodal treatment in supplementary or standalone prescription or nonprescription software-based digital therapeutics (PDT/DTx), being developed by Click Therapeutics, Inc.

DETAILED DESCRIPTION:
CT-100 is a platform that provides an interactive, software based therapeutic component (CT-100-001) that may be used as part of a multimodal treatment in future prescription or non-prescription software-based digital therapeutics (PDT/DTx). CT-100-001 contains a class of Digital Neuro-activation and Modulation (DiNaMo) component. This DiNaMo component targets key neural systems (including, but not limited to, systems related to cognitive control, sensory-, perceptual-, affective-, pain-, attention-, social-, and self-processing) to optimally improve patients' cognitive and mental health. The CT-100-001 DiNaMo component is designed to improve cognitive impairments and mood challenges.

The purpose of the proposed basket study is to evaluate the initial effects of the CT-100-001, a DiNaMo component (the Study App) on cognitive functioning and related outcomes compared to Care-As-Usual across several non-DSM-5 indications. These indications have known high prevalence of cognitive impairments due to the illness and/or treatments. such as in Multiple Sclerosis, Breast or Lung Cancer, and Mild Cognitive Impairment.

ELIGIBILITY:
Inclusion Criteria:

A participant will be eligible for entry into the study if all the following criteria are met:

1. Age ranges in years: 22-52 for Multiple Sclerosis, 35-65 for Cancer (Breast or Lung), and 45-75 for Mild Cognitive Impairment.
2. Diagnosis of indication under study (Multiple Sclerosis, Cancer - Breast or Lung, Mild Cognitive Impairment)
3. Self-reported cognitive impairment and mood symptoms that began in the context of the primary indication under study.
4. Fluent in written and spoken English (confirmed by ability to read and comprehend the informed consent form.)
5. Willing and able to comply with study protocol and assessments, evidenced by completion of the Screening Survey.
6. Lives in the United States.
7. Has an active email address and is willing and able to receive email messages.
8. Is the sole user of an iPhone or a smartphone with an Android operating system, and with cellular and/or internet access for the duration of the study period.

Exclusion Criteria:

A participant is excluded from the study if any of the following criteria apply:

1. Physician-diagnosed insomnia in the Screening Survey.
2. Cognitive impairment/mood symptoms or clinical diagnosis of depression attributed to a condition other than the underlying medical condition.
3. Is currently pregnant or breastfeeding.
4. Substance use disorder within the past 1 year.
5. Initiation or change in central nervous system-active medication (e.g., antidepressants) during the last 2 months.
6. Participation in a clinical trial within the last 3 months.
7. Anticipates a lifestyle change or change in current treatment during the study period that could affect cognitive functioning.
8. Visual, dexterity or cognitive deficit so severe that precludes the use of an app.
9. Severe neurological disorders impairing brain function.
10. Psychiatric hospitalization in the past 6 months.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
PROMIS Item Bank v2.0 - Cognitive Function - Short Form 8a (PROMIS-CF) | Baseline (Day 1) corrected change of intervention vs, Care-As-Usual on Day 21
  Change in cognitive functioning as measured by PROMIS Item Bank v2.0 - Cognitive Function - Short Form 8a (PROMIS-CF) in the Study App intervention group compared to a Care-As-Usual control group; 8 items, from minimum of 8 (worst) to maximum of 40 (best)

SECONDARY OUTCOMES:
Patient-reported Quality-of-Life (QoL) as measured by the PROMIS-29 in the Study App intervention group compared to a Care-As-Usual control group | Baseline (Day 1) corrected change of intervention vs, Care-As-Usual on Day 21
  To explore changes in patient-reported Quality-of-Life (QoL) as measured by the PROMIS-29 in the Study App intervention group compared to a Care-As-Usual control group; 29 items across mood (2 domains), physical function, pain interference, fatigue, sleep disturbance, ability to participate in social roles and activities and cognitive function on a scale of 1 (worst) to 5 (best), and pain intensity (on a scale ranging from 0 (no pain) to 10 (worst pain imaginable).
Global Rating of Change (GRC-Cognition and GRC-Mood) | Baseline (Day 1) corrected change of intervention vs, Care-As-Usual on Day 21
  Treatment impact reported at week 3 as measured by Global Rating of Change (GRC-Cognition and GRC-Mood) in the Study App intervention group compared to a Care-As-Usual control group; -5 (worst), 0 unchanged, 5 (best - recovered)
Changes in indication-specific measures of Symbol Digit Modalities Test (SDMT) in Multiple Sclerosis (only) | Baseline (Day 1) corrected change of intervention vs, Care-As-Usual on Day 21
  To explore changes in indication-specific measures of Symbol Digit Modalities Test (SDMT) in the Study App intervention group compared to a Care-As-Usual control group in in Multiple Sclerosis.
  For SDMT, scoring involves summing the number of correct substitutions within the 90 second interval, minimum: 0 (worst), max: 110 (best).
Changes in indication-specific measures of Functional Assessment of Cancer Therapy-Cognitive (FACT-Cog) in Cancer (Breast/Lung; only). | Baseline (Day 1) corrected change of intervention vs. Care-As-Usual on Day 21
  To explore changes in indication-specific measures of Functional Assessment of Cancer Therapy-Cognitive (FACT-Cog) in the Study App intervention group compared to a Care-As-Usual control group in Cancer (Breast/Lung).
  For FACT-Cog, scoring involves 37-item Likert-scaled questionnaire with responses ranging from 0 to 4 and consisting of four subscales (Perceived Cognitive Impairments, Perceived Cognitive Abilities, Impact on Quality Of Life, Comments From Others). Higher scores are better (better functioning or quality of life): minimum 0 (worst), maximum 4 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Lakhan, MDPhD, FAAN, Study Director — Click Therapeutics; Jacqueline Lutz, PhD, Study Director — Click Therapeutics
Locations (1):
- Click Therapeutics, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No